CLINICAL TRIAL: NCT02613455
Title: Prospective Randomize Trial Comparing Corticosteroid Injection to High Energy Extracorporeal Shock Wave Therapy for Lateral Epicondylitis
Brief Title: Corticosteroid Injection Verses High Energy Extracorporeal Shock Wave Therapy for Lateral Epicondylitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 405072-2
Record Dates: First submitted 2015-10-28; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Triamcinolone Acetonide; Triamcinolone; Adrenal Cortex Hormones; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kenalog (triamcinolone ) (Active Comparator): Patients assigned to the corticosteroid arm will receive an intratendinous injection of 1cc Kenalog-40 (triamcinolone-40mg) + 2cc lidocaine 1% by an attending orthopaedic hand surgeon in clinic. They will be provided a home stretching regimen for lateral epicondylitis. They will be discouraged from using nonsteroidal anti-inflammatory drugs . No additional physical or occupational therapy will prescribed.
  Interventions: Drug: Kenalog (triamcinolone); Drug: lidocaine 1% (lidocaine HCl 20mg)
- extracorporeal shock wave therapy (Active Comparator): Following clearance, patients will be booked for ESWT in the operating room either Walter Reed National Military Medical Center (WRNMMC) or Kimbrough Ambulatory Care Center (KACC), depending on availability. Under conscious sedation, patients will receive 2000 shocks at 18-24 kilovolts, which is the standard dose utilized by our clinic in treatment of this condition. The range is necessary to account for differing size of the soft tissue envelope depending on patient habitus. The final dose utilized will be at the surgeon's discretion.
  Interventions: Procedure: extracorporeal shock wave therapy

INTERVENTIONS:
Procedure: extracorporeal shock wave therapy — Following clearance, patients will be booked for ESWT in the operating room either WRNMMC or Kimbrough Ambulatory Care Center (KACC), depending on availability. Under conscious sedation, patients will receive 2000 shocks at 18-24kV, which is the standard dose utilized by our clinic in treatment of this condition. The range is necessary to account for differing size of the soft tissue envelope depending on patient habitus. The final dose utilized will be at the surgeon's discretion.
  Other Names: ESWT
  Arms: extracorporeal shock wave therapy
Drug: Kenalog (triamcinolone) — patients will receive an intratendinous injection in the common tendon origin of the extensor/supinators at the lateral epicondyle by an attending orthopaedic hand surgeon. The injection will contain 1cc of Kenalog-40 (triamcinolone 40mg) + 2cc lidocaine 1% (lidocaine HCl 20mg). This is the standard dose for lateral epicondylitis used routinely in the WRNMMC orthopaedic clinic.
  Other Names: Steriod, Corticosteroid
  Arms: Kenalog (triamcinolone )
Drug: lidocaine 1% (lidocaine HCl 20mg) — patients will receive an intratendinous injection in the common tendon origin of the extensor/supinators at the lateral epicondyle by an attending orthopaedic hand surgeon. The injection will contain 1cc of Kenalog-40 (triamcinolone 40mg) + 2cc lidocaine 1% (lidocaine HCl 20mg). This is the standard dose for lateral epicondylitis used routinely in the WRNMMC orthopaedic clinic.
  Other Names: lidocaine
  Arms: Kenalog (triamcinolone )

SUMMARY:
The purpose of this study is to prospectively compare the pain and functional outcomes of patients with chronic lateral epicondylitis treated with either intratendinous corticosteroid injection or high energy extracorporeal shock wave therapy (ESWT).

DETAILED DESCRIPTION:
Corticosteroid injections and high energy ESWT are standard therapies for lateral epicondylitis at Walter Reed National Military Medical Center. While corticosteroid injections have been shown to be moderately effective in the short term for the condition, a significant minority of patients remains symptomatic. Low energy ESWT has mixed results in the orthopaedic literature, but to date no study has specifically examined the effects of high energy ESWT. The investigators plan to randomize a total of 80 patients with the diagnosis of lateral epicondylitis to either corticosteroid injection or high energy ESWT, and follow them for a total of 12 months. Primary outcomes will be Disabilities of the Arm, Shoulder, and Hand (DASH) score, Patient Reported Tennis Elbow Evaluation (PRTEE) score, Mayo Elbow Score, Veterans Rand-36, and return-to-work status. Patients will be surveyed at baseline, 6 weeks, 3 months, and 6 months. All assessments will be done by an independent physician examiner who is blinded to the treatment received.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the WRNMMC orthopaedic hand surgery clinic for complaints of lateral elbow pain will be evaluated for inclusion in the study. Inclusions criteria will be:
* Clinical diagnosis of lateral epicondylitis based on primary complaint of lateral elbow pain and either (a) tenderness over the lateral epicondyle with direct palpation, or (b) exacerbation of pain at the lateral elbow with resisted dorsiflexion of the wrist
* Failure of previous trial of non-operative management of at least 4wks duration (to include rest/light duty, non steroidal anti-inflammatory drugs , physical/occupational therapy, home stretching regimen)

Exclusion Criteria:

* Age <18yo
* Pregnant or planning to become pregnant during study period (based on verbal questioning)
* Steroid treatment (oral or injectable) within the previous 3mo
* Diagnosis of ipsilateral compressive neuropathy
* Allergy to Kenalog, lidocaine, or conductive ultrasound gel
* Diagnosis of inflammatory arthropathy or rheumatoid conditions
* Diagnosis of fibromyalgia, chronic fatigue syndrome, complex regional pain syndrome, or other chronic widespread pain syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6 months
  VAS is a measurement instrument to quantify pain. Difference between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy at six months following intervention.
Disabilities of the Arm, Shoulder and Hand (DASH) | 6 months
  DASH is a questionnaire to measure upper extremity symptoms and ability to perform activities. Difference between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy at six months following intervention.
Mayo Elbow Score | 6 months
  Mayo Elbow score is an elbow focused outcome score. Difference between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy at six months following intervention.
Veteran Rand 36 Item Health Survey (VR-36) | 6 months
  VR-36 is a 36 item health survey widely used in the veteran population. Difference between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy at six months following intervention.
Patient-Related Tennis Elbow Evaluation (PRTEE) | 6 months
  PRTEE is a questionnaire to measure pain and disability in patients with lateral epicondylitis. Difference between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy at six months following intervention.

SECONDARY OUTCOMES:
Grip Strength | 6 months
  Difference in grip strength between the Kenalog (triamcinolone ) group and extracorporeal shock wave therapy will be determined at six months following intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Tintle, MD, Principal Investigator — WRNMMC Orthopaedics
Locations (1):
- Walter Reed National Military Medical Ceneter, Bethesda, Maryland, United States